CLINICAL TRIAL: NCT04199208
Title: The Effect of Prehabilitation on Surgical Complications Following Colon Surgery - a Prospective Randomized Study
Brief Title: Does Prehabilitation Improve Outcome in Coloncancer Surgery?
Acronym: PRIO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRIO01
Record Dates: First submitted 2019-12-09; First posted 2019-12-13 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Surgery--Complications
Keywords: exercise therapy; perioperative period; coloncancer
MeSH Terms: interventions — Preoperative Exercise; Immunonutrition Diet

STUDY DESIGN:
Intervention Model Description: Randomized two-armed clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Arm (Active Comparator): Standard perioperative care is given.
  Interventions: Other: Standard Care Arm
- Interventional Arm (Experimental): Intervention of prehabilitation and immunonutrition is given prior to surgery
  Interventions: Other: Prehabilitation and Immunonutrition

INTERVENTIONS:
Other: Prehabilitation and Immunonutrition — See study synopsis
  Arms: Interventional Arm
Other: Standard Care Arm — Standard care as per the daily routines of the Hospital at which the study takes place
  Arms: Standard Care Arm

SUMMARY:
The study aims to find out if complications after surgery for large bowel (colon) cancer can be reduced or avoided in the most frail and elderly by letting them go through an exercise- and diet regime prior to the surgical procedure.

DETAILED DESCRIPTION:
All patients with colon cancer who are intended for curative surgery without neoadjuvant chemotherapy who are >=60 years old will be screened with an ergospirometry. The ones that have a ventilate anaerobic threshold (VAT) of less than 11 mg/ml/kg will be included in the study as they are considered extra frail and have a previously proven high risk for complications. These patients will be randomized to standard care or an intervention of prehabilitation consisting of immunonutrition (protein supplement, multivitamin supplement, Selene etc) and an exercise regimen with 4x1 hours per week of cycling on an ergometer. The exercise regimen will be performed in a group of patients and will be led by a physical therapist to ensure compliance. The resistance of the ergometer will be standardized according to the patient's VAT.

The primary outcome measures will be number of and severity of postoperative complications. Secondary outcome measures include quality of life during prehabilitation with repeated measurements during 5 years after surgery, disease-free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of older
* Colon cancer diagnosis (macroscopic, microscopic or x-ray diagnosed)
* Ventilatory Anaerobic Threshold <11mg/ml/kg
* Planned open or laparoscopic colectomy due to colon cancer

Exclusion Criteria:

* Lower extremity amputee
* Disease requiring radio- and/or chemotherapy prior to surgery/palliative disease
* Distal metastases (Locoregional lymph nodes are OK)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2023-01-07 (Estimated); Study Completion 2028-01-07 (Estimated)

PRIMARY OUTCOMES:
Complications | Assessed when patient is discharged from hospital
  Severity of postoperative complications according do Clavien-Dindo
Complications | Assessed at postoperative day 5.
  Number of complication(s) according to POMS

SECONDARY OUTCOMES:
Quality of life with SF-36 | At point in time when patient is informed of the cancer, after prehabilitation (just before surgery), 30 days, 2, 3 and 6 months, 1, 3 and 5 years after surgery.
  Quality of life
Disease-free survival | 30 and 90 days after surgery, 1, 3 and 5 years after surgery.
  Cancer-free survival Cancer-free survival of the group of the group
Overall survival | 30 and 90 days after surgery, 1, 3 and 5 years after surgery.
  Overall survival of the group (taking all causes of death into account)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Öberg, MD, PhD, Principal Investigator — Region Skåne/Lund University

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT04199208/Prot_SAP_000.pdf